CLINICAL TRIAL: NCT02010099
Title: A Prospective, Randomized, Three Arms, Open Label Study Comparing the Safety and Efficacy of Two Formulations of PP110 to the Active Comparator Preparation-H® Cream in the Treatment of Bleeding Hemorrhoids Grades 2-3
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peritech Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP110 01
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Bleeding Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PP110 Gel (Experimental): PP110 Gel
  Interventions: Drug: PP110 Gel
- PP110 medicated wipes (Experimental): PP110 Medicated wipes
  Interventions: Drug: PP110 Medicated wipes
- Preparation-H cream (Active Comparator): Preparation-H cream
  Interventions: Drug: Preparation-H Cream

INTERVENTIONS:
Drug: PP110 Gel
  Arms: PP110 Gel
Drug: PP110 Medicated wipes
  Arms: PP110 medicated wipes
Drug: Preparation-H Cream
  Arms: Preparation-H cream

SUMMARY:
Eligible patients with bleeding hemorrhoids of grade 2-3 are randomized to test-1 product (PP110 Gel), test-2 product (PP-110 medicated wipes) or control (Preparation-H cream).

Test product usage: once daily, about 1-5 minutes prior to first bowel movement. Control product usage: according to label, 3-4 times daily application to rectal region.

At the end of each day, subject fills a questionnaire regarding bleeding, pain, discharge, swelling, itching, discomfort and painkiller usage.

Treatment is for two weeks, after which subjects fill a feedback questionnaire addressing treatment efficacy and subject satisfaction. Also, at the end of two weeks, subjects are examined by study physician who assesses hemorrhoid severity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70
2. Bleeding hemorrhoids with / without pain
3. Diagnosis of internal hemorrhoids of grade 2-3, or external bleeding hemorrhoids
4. Signed Informed Consent

Exclusion Criteria:

1. Known rectal sensitivity
2. Rectal infection
3. Grade IV hemorrhoids
4. Use of anti-coagulants (except Aspirin or Plavix) within 30 days prior to enrollment
5. Known inflammatory bowel disease
6. Anal fissure
7. Military personnel
8. Female patients that are pregnant, or are not using a reliable method of birth control, or are nursing
9. Patients who have been involved in another experimental trial within the past 30 days
10. Patients presently diagnosed with cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Bleeding / Spotting | 14 days

SECONDARY OUTCOMES:
Pain | 14 days
Discharge | 14 days
Itching | 14 days
Swelling | 14 days
Discomfort | 14 days
Painkillers usage | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Klein, Prof., Principal Investigator — Maccabi Healthcare Services, Israel
Locations (5):
- Israel (5):
  - Kfar Saba
  - Kiryat Ono
  - Modiin
  - Ramat Gan
  - Tel Aviv